CLINICAL TRIAL: NCT02013648
Title: Randomized Phase III Study of Intensive Chemotherapy With or Without Dasatinib (Sprycel™) in Adult Patients With Newly Diagnosed Core-Binding Factor Acute Myeloid Leukemia (CBF-AML)
Brief Title: Randomized Phase III Study of Intensive Chemotherapy With or Without Dasatinib (Sprycel™)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Prof. Dr. Hartmut Doehner, Prof. Dr., University of Ulm
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMLSG 21-13
Record Dates: First submitted 2013-12-11; First posted 2013-12-17 (Estimated); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Acute Myeloid Leukemia (AML)
Keywords: AML; Dasatinib; Core Binding Factor (CBF)
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Dasatinib; Cytarabine; Daunorubicin; Idarubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard arm (Active Comparator): Patients will receive induction therapy with daunorubicin 60 mg/m2/day administered on days 1-3 (when daunorubicin is not available due to supply shortage: Idarubicin 12mg²/day on days 1,3,5) and cytarabine 200 mg/m2/day administered by continuous IV infusion on days 1-7.
  Patients achieving PR only at the end of cycle 1 will receive a second induction cycle with daunorubicin 50 mg/m2/day (when daunorubicin is not available due to supply shortage: Idarubicin 10 mg²/day on days 1 and 3) administered on days 1-3 and cytarabine 200 mg/m2/day administered by cont. IV infusion daily on days 1-5.
  Patients will receive 4 cycles of consolidation therapy. Consolidation therapy consists of high-dose cytarabine 3 g/m2 (>60 years: 1 g/m2) q12h, days 1-3 administered intravenously over three hours.
  Follow-up period: There is no maintenance therapy in the standard arm. Patients will be closely followed, in particular for molecular disease persistence or molecular relapse.
  Interventions: Drug: Cytarabine; Drug: Daunorubicin; Drug: Idarubicin
- Investigational arm (Experimental): Patients will receive induction therapy with daunorubicin 60 mg/m2/day on days 1-3 (when daunorubicin is not available due to supply shortage: Idarubicin 12mg²/day on days 1,3,5) and cytarabine 200 mg/m2/day by cont. IV infusion on days 1-7. Patients will receive dasatinib 100 mg QD on days 8-21. Patients achieving PR only at the end of cycle 1 will receive a 2nd induction cycle with daunorubicin 50 mg/m2/day on days 1-3 (when daunorubicin is not available due to supply shortage: Idarubicin 10 mg²/day on days 1 and 3) and cytarabine 200 mg/m2/day by cont. IV infusion on days 1-5. Patients will receive dasatinib 100 mg QD on days 6-21.
  Consolidation therapy (4 cycles). Treatment consists of high-dose cytarabine 3 g/m2 (>60 years: 1 g/m2) q12h, days 1-3 iv over 3 hours. Patients will receive dasatinib 100 mg QD on days 4-21. Maintenance therapy: Patients completing consolidation therapy will continue to receive single agent dasatinib 100 mg QD for one year (or until relapse).
  Interventions: Drug: Dasatinib; Drug: Cytarabine; Drug: Daunorubicin; Drug: Idarubicin

INTERVENTIONS:
Drug: Dasatinib
  Other Names: Sprycel
  Arms: Investigational arm
Drug: Cytarabine
  Other Names: ARA-cell
Drug: Daunorubicin
  Other Names: Daunoblastin
Drug: Idarubicin

SUMMARY:
This is a randomized phase III open-label, multicenter trial evaluating standard induction therapy (daunorubicin [DNR] and cytarabine [Ara-C]) and consolidation therapy (high-dose cytarabine [HDAC]) with or without dasatinib in adult patients with newly diagnosed CBF-AML

DETAILED DESCRIPTION:
This is a randomized phase III open-label, multicenter trial evaluating standard induction therapy (daunorubicin [DNR] and cytarabine [Ara-C]) and consolidation therapy (high-dose cytarabine [HDAC]) with or without dasatinib in adult patients with newly diagnosed CBF-AML; in the investigational arm, consolidation therapy is followed by a one-year maintenance therapy with dasatinib. Patients with molecular disease persistence or molecular relapse as assessed by quantitative RQ-PCR for the CBF fusion transcripts will be eligible for hematopoietic stem cell transplantation before overt hematologic relapse occurs. Primary endpoint is event-free survival.

AML patients will be assessed for the CBF fusion genes in one of two AMLSG central laboratories within 48 hours of diagnosis, and only patients with CBF-AML will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Core-binding factor (CBF) AML with molecular diagnosis of RUNX1-RUNX1T1 fusion transcript resulting from t(8;21)(q22;q22.1) (or a variant form) or of CBFB-MYH11 fusion transcript resulting from inv(16)(p13.1q22)/t(16;16)(p13.1;q22) as assessed in one of the central AMLSG reference laboratories (Ulm, Hannover)
* Age ≥ 18; there is no upper age limit
* No prior chemotherapy for leukemia except hydroxyurea for up to 5 days during the diagnostic screening phase
* Non-pregnant and non-nursing. Due to the unknown teratogenic potential of dasatinib in humans, pregnant or nursing patients may not be enrolled. Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test within a sensitivity of at least 25 mIU/mL with-in 72 hours prior to registration. Women of child-bearing potential must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control - one highly effective method (e.g., IUD, hormonal, tubal ligation, or partner's vasectomy), and one additional effective method (e.g., latex condom, diaphragm, or cervical cap) - AT THE SAME TIME, at least four weeks before she begins dasatinib therapy. "Women of childbearing potential" is defined as a sexually active mature woman who has not undergone a hysterectomy or who has had menses at any time in the preceding 24 consecutive months.
* Men must agree not to father a child and must use a latex condom during any sexual contact with women of childbearing potential while taking dasatinib and for 3 months after therapy is stopped, even if they have undergone a successful vasectomy.
* Signed written informed consent.

Exclusion Criteria:

* Performance status WHO >2
* Pulmonary edema and/or pleural/pericardial effusion within 14 days of day 1. If edema/effusion resolves to CTC Grade ≤1, patients can be treated with dasatinib.
* Patients with ejection fraction <50% by echocardiography within 14 days of day 1
* Organ insufficiency (creatinine >1.5x upper normal serum level; bilirubin, AST or AP >2.5x upper normal serum level; heart failure NYHA III/IV; severe obstructive or restrictive ventilation disorder)
* Uncontrolled infection
* Patients with a "currently active" second malignancy other than non-melanoma skin cancers. Patients are not considered to have a "currently active" malignancy, if they have completed therapy and are considered by their physician to be at less than 30% risk of relapse within one year.
* Severe neurological or psychiatric disorder interfering with ability of giving an informed consent
* Known positive for HIV, active HBV, HCV, or Hepatitis A infection
* Bleeding disorder independent of leukemia
* No consent for registration, storage and processing of the individual disease characteristics and course as well as information of the family physician and/or other physicians involved in the treatment of the patient about study participation.
* No consent for biobanking.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2014-07; Primary Completion 2024-02 (Actual); Study Completion 2024-02 (Actual)

PRIMARY OUTCOMES:
Event-free Survival | 4 years
  To assess event-free survival (EFS) after intensive induction (daunorubicin and cytarabine) and consolidation (high-dose cytarabine) chemotherapy with or without dasatinib in patients with CBF-AML

SECONDARY OUTCOMES:
Cumulative incidence of relapse (CIR) | 4 years
Cumulative incidence of death (CID) | 4 years
overall survival | 4 years
relapse-free survival | 4 years
PIA analysis | 4 years
  Pharmacodynamic inhibition of KIT as assessed by the KIT plasma inhibitory assay (PIA)
toxicity | 7 months (standard arm) / 19 months (investigational arm)
  Type, frequency, severity (graded using the National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] version 4.03), timing and relatedness of non-hematologic toxicity observed during different treatment cycles.

CONTACTS AND LOCATIONS:
Overall Officials: Hartmut Doehner, Prof. Dr., Principal Investigator — University of Ulm
Locations (54):
- Austria (5):
  - Universitätsklinik für Innere Medizin V, Innsbruck
  - Krankenhaus der Barmherzigen Schwestern, Linz
  - Krankenhaus der Elisabethinen Linz GmbH, Linz
  - Universitätsklinik der PMU, Salzburg
  - Hanuschkrankenhaus, Vienna
- Germany (49):
  - MVZ Osthessen, Fulda, Hesse
  - Universitätsklinikum Schleswig-Holstein, Kiel, Schleswig-Holstein
  - Klinikum Aschaffenburg-Alzenau, Aschaffenburg
  - Helios Klinikum Bad Saarow, Klinik für Hämatologie, Bad Saarow
  - Klinikum am Urban, Berlin
  - Klinikum Neukölln, Berlin
  - Charité Universitätsmedizin Campus Virchow Klinikum, Berlin
  - Knappschaftskrankenhaus Bochum, Bochum
  - Universitätsklinikum Medizinische Klinik und Poliklinik III, Bonn
  - Städtisches Klinikum Braunschweig gGmbH, Braunschweig
  - Klinikum Bremen Mitte gGmbH, Bremen
  - Klinikum Darmstadt Medizinische Klinik V, Darmstadt
  - St. Johannes Hospital, Dortmund
  - Universitätsklinikum Medizinische Klinik und Poliklinik, Düsseldorf
  - Klinikum Esslingen, Esslingen am Neckar
  - Malteser Krankenhaus St. Franziskus-Hospital, Flensburg
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Wilhelm-Anton-Hospital gGmbH, Goch
  - Universitätsmedizin Göttingen, Göttingen
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Klinikum Hanau GmbH, Hanau
  - Klinikum Region Hannover GmbH, Hanover
  - Medizinische Hochschule Hannover, Hanover
  - SLK-Kliniken GmbH, Heilbronn
  - Marienhospital Klinikum der Ruhr-Universität, Herne
  - Universitätsklinikum des Saarlandes, Homburg
  - Städtisches Klinikum Karlsruhe gGmbH, Karlsruhe
  - Gemeinschaftspraxis Hämato-Onkologie, Lebach
  - Klinikum Lippe GmbH, Lemgo
  - Märkische Kliniken GmbH, Lüdenscheid
  - Univ-Klinikum der Otto-von Guericke-Universität, Magdeburg
  - III. Medizinische Klinik und Poliklinik Universitätsmedizin der Johannes Gutenberg-Universität, Mainz
  - Johannes Wesling Klinikum, Minden
  - Stauferklinikum Schwäbisch Gmünd, Mutlangen
  - Klinikum rechts der Isar der TU, München
  - Ortenau Klinikum, Offenburg
  - PIUS Hospital, Oldenburg
  - Klinikum Oldenburg gGmbH, Oldenburg
  - Klinikum Passau, Passau
  - Universitätsklinikum Regensburg, Regensburg
  - Caritasklinkum Saarbrücken St. Theresia, Saarbrücken
  - Klinikum Stuttgart, Stuttgart
  - Vinzenz von Paul Kliniken gGmbH Marienhospital, Stuttgart
  - Klinikum Mutterhaus der Borromäerinnen gGmbH, Trier
  - Medizinische Universitätsklinik, Tübingen
  - Universitätsklinikum Ulm Zentrum für Innere Medizin, Ulm
  - Schwarzwald-Baar Klinikum, Villingen-Schwenningen
  - Kliniken Essen Süd, Werden
  - HELIOS Klinikum, Wuppertal

REFERENCES:
- [Derived] Dohner H, Spath D, Saadati M, Fiedler W, Gotze KS, Koller E, Westermann J, Vogel W, Heuser M, Lubbert M, Tischler HJ, Germing U, Teichmann LL, Fransecky L, Wolfler A, Nachbaur D, Hertenstein B, Schroers R, Martens UM, von Harsdorf S, Radsak MP, Aschauer G, Weisshaar S, Corbacioglu A, Schrade A, Gaidzik VI, Thol FR, Paschka P, Bullinger L, Benner A, Dohner K, Ganser A. Phase 3 study of intensive chemotherapy with or without dasatinib in core-binding factor acute myeloid leukemia. Blood. 2026 Jan 5:blood.2025030722. doi: 10.1182/blood.2025030722. Online ahead of print. PMID 41490515
- [Derived] Paschka P, Schlenk RF, Weber D, Benner A, Bullinger L, Heuser M, Gaidzik VI, Thol F, Agrawal M, Teleanu V, Lubbert M, Fiedler W, Radsak M, Krauter J, Horst HA, Greil R, Mayer K, Kundgen A, Martens U, Heil G, Salih HR, Hertenstein B, Schwanen C, Wulf G, Lange E, Pfreundschuh M, Ringhoffer M, Girschikofsky M, Heinicke T, Kraemer D, Gohring G, Ganser A, Dohner K, Dohner H. Adding dasatinib to intensive treatment in core-binding factor acute myeloid leukemia-results of the AMLSG 11-08 trial. Leukemia. 2018 Jul;32(7):1621-1630. doi: 10.1038/s41375-018-0129-6. Epub 2018 Apr 17. PMID 29720733